CLINICAL TRIAL: NCT04993794
Title: Additive Anti-inflammatory Action for Critically Ill Patients With Cardiovascular Surgery (Xuebijing) IV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5A-Plan IV
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Disease; Aortic Dissection; Coronary Artery Disease; Valve Heart Disease; Congenital Heart Disease; Critical Illness
MeSH Terms: conditions — Cardiovascular Diseases; Aortic Dissection; Coronary Artery Disease; Heart Valve Diseases; Heart Defects, Congenital; Critical Illness | interventions — Xuebijing; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XueBiJing (Active Comparator): XBJ (Composed of Carthamus tinctorius L., Paeonia Lactifora Pall, Ligusticum wallichii, Salvia miltiorrhiza, Angelica sinensis, etc. Tianjin Chase Sun Pharmaceutical Group, Tianjin, China, batch No. 1603231) 100ml Xuebijing injection every 12 h (q12h) for 60 min
  Interventions: Drug: XueBiJing Injection
- Normal saline (Placebo Comparator): 0.9% saline every 12 h (q12h) for 60 min
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: XueBiJing Injection — XueBiJing, specification 10mL/ampule, packaging 10 ampules/container, concentration 0.1g/mL, were manufactured by a Good Manufacturing Practice certified company in China (Tianjin Chase Sun Pharmaceutical Co., Tianjin, China; China lot number 1304291, 1401091 and, 1501261). Generally, the treatment duration of the study was at least 5 days.
  Arms: XueBiJing
Drug: Normal saline — Same saline dose as XueBiJing injection is taken intravenously.
  Arms: Normal saline

SUMMARY:
XueBiJing, a Chinese herbal derived therapeutic, has been approved to treat severe infections (sepsis) in critically ill patients (China Food and Drug Administration; Beijing, China, Number Z20040033). Cardiopulmonary bypass (CPB) will produce large amounts of inflammatory mediators and oxygen free radicals, which causes the lipid peroxidation damage and mononuclear cell migration, thus aggravating organ inflammation and damage. Therefore, exploring new methods to prevent and alleviate organ injury caused by CPB is an important topi in clinical practice. However, little knowledge is regarding the effect of Xuebijing injection on CPB-related organ injury. To answer these questions, the authors conducted this randomized trial to compare XueBiJing with placebo in critically ill patients with cardiovascular surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received cardiovascular surgery fulfilled three or more of the following criteria:

   * Pao2/Fio2 ratio less than or equal to 250mm Hg,
   * Respiratory rate greater than or equal to 30 breaths/min,
   * Blood urea nitrogen greater than 20mg/dL,
   * WBC count < 4,000 cells/mm3 or >15 000 cells/mm3 not due to other causes,
   * Core temperature < 36°C or >38.5°C,
   * Receiving treatment with vasopressors at therapeutic doses after adequate fluid resuscitation,
   * radiographic findings of new pulmonary infiltrate(s).
2. Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Pregnant and lactating women.
2. Allergic to Xuebijing and its ingredients, or have severe allergies.
3. Mental illness with poor compliance.
4. Severe primary disease (active pulmonary tuberculosis, asthma, cystic pulmonary fibrosis, pulmonary sarcoidosis, pulmonary interstitial fibrosis, unresectable tumors, blood diseases, Alzheimer s disease, or HIV).
5. Participation in other clinical trials in the previous 30 days.
6. Patients who are unsuitable for participation or unable to participate in this trial according to the judgment of the investigators (existing risk of potential medical disputes, and severe heart failure limiting the amount of liquid intake).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | up to 30 days after surgery

SECONDARY OUTCOMES:
Highest Sequential Organ Failure Assessment score | 7 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of nanjing medical university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided